CLINICAL TRIAL: NCT00361972
Title: Elucidation of Acid-Induced Pulmonary Inflammation
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: limited recruitment
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kathryn A. Peterson, md, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15444; IRB #15444
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-06

CONDITIONS: Gastroesophageal Reflux; Asthma
MeSH Terms: conditions — Gastroesophageal Reflux; Asthma | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lansoprazole therapy (Active Comparator): Lansoprazole 30 mg orally twice daily
  Interventions: Drug: lansoprazole
- Placebo (Placebo Comparator): placebo orally twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lansoprazole — 30 mg of lansoprazole twice daily for 6 weeks
  Other Names: Prevacid
  Arms: Lansoprazole therapy
Drug: placebo — placebo comparator to lansoprazole 30 mg, twice daily for 6 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate how heartburn may lead to different types of inflammation in one's airways. Additionally, the study will determine whether aggressive treatment of heartburn results in improvement in both symptoms of heartburn and asthma but also in documented improvement in airway inflammation as determined by biopsy. The results of this study will be important in directing future research into the relationship between heartburn and asthma and may provide a clue whether certain subtypes of asthma may be caused primarily by gastroesophageal reflux (GER).

DETAILED DESCRIPTION:
Currently, many Americans suffer from asthma. The exact mechanism by which airway inflammation leads to asthma symptoms has yet to be clearly explained. In previous studies, persons with asthma appear to have different types of inflammation in their lungs. The reasons for this difference remain a mystery. Allergy is known to play a role in bronchospasm. Other mechanisms have not been discovered.

It is known that asthma and heartburn are correlated. Studies have confirmed a direct relationship between cough and heartburn (Gastroesophageal reflux). Other researchers have determined that asthma is often worsened by GER. Determination of the exact relationship between these two entities remains unclear.

Heartburn may contribute to airway inflammation in asthmatics, resulting in different patterns of inflammation between those people with and without GER. In fact, adult-onset asthma may result primarily from longstanding heartburn. This has yet to be proven.

This study will evaluate how heartburn may lead to different types of inflammation in one's airways. Additionally, the goal of this study is to determine whether aggressive treatment of heartburn results in improvement in both symptoms of heartburn and asthma but also in documented improvement in airway inflammation as determined by biopsy. The results of this study will be important in directing future research into the relationship between heartburn and asthma and may provide a clue whether certain subtypes of asthma may be caused primarily by GER.

A total of 30 subjects will be studied, randomized to twice daily lansoprazole or placebo. Study procedures are as follows:

A. Esophageal studies and validated questionnaires:

Patients will be evaluated with validated SF-36 Quality of Life Questionnaire, Mini-asthma Quality of Life Questionnaire, and GER Questionnaire. Patients will undergo esophageal manometry and pH detection with a 24- hour pH probe to confirm the presence of pathologic GER.

B. Bronchoscopy:

After an overnight fast, subjects will report to the bronchoscopy suite as directed. Bronchoscopy with bronchoalveolar lavage (BAL) and bronchial biopsy will be performed following the University of Utah's standardized protocol. Bronchoscopy and endobronchial biopsies present minimal risk to asthmatic airways when performed by appropriate, trained personnel. Conscious sedation with intravenous remifentanyl and propofol will be administered by a trained nurse experienced in conscious sedation. The nose and pharynx will be anesthetized with 1% lidocaine administered by nebulization and by lidocaine jelly administered topically to the nasal mucosa. Additional lidocaine will be administered via the bronchoscope to the vocal cords, trachea, main carina and mainstem bronchi. The total dose of lidocaine will not exceed 400 mg. All subjects will have continuous cardiac and oxygen saturation monitoring and will receive supplemental oxygen during the procedure sufficient to maintain SpO2 > 90%.

The subject will be placed in a recumbent position and the bronchoscope will be introduced via the nose. After passing the vocal cords, the bronchoscope will be introduced via the right mainstem bronchus into the right middle lobe where it will be wedged into a segmental bronchus. (Should, for any reason, the right middle lobe be inaccessible, the same procedure will be used to wedge the bronchoscope into a lingular segment in the left lung.) A 60 cc aliquot of room temperature normal saline will be instilled through the bronchoscope and recovered using the same syringe. This procedure will be repeated three more times (total lavage volume of 240 cc) and the recovered volumes will be pooled and measured. Forceps biopsies of respiratory mucosa will then be taken from the trachea, main carina, bronchus intermedius and right middle lobe areas. Two to six biopsies will be taken from each site. Specific tissue from each site will be frozen and stored for future use.

Individuals will be randomized to lansoprazole 30 mg twice daily or placebo (all patients will undergo lifestyle modification for reflux) for 6 weeks. It has been determined in previous studies that higher levels of acid suppression are needed to result in clinical improvement in asthma.

Patients will be monitored by telephone at regular intervals. Rescue inhaler use, hospitalizations, exercise tolerance, and study compliance will be assessed and recorded to document clinical progress. Patients will be asked to maintain their standard inhaler therapy (especially that of inhaled steroids). Any changes to the therapy will be immediately reported to the investigators. If subjects experience an acute flare, appropriate medications will be given until the patient is stable to return to their initial inhaler regimen. If patients remain on stable medication throughout the trial, repeat bronchoscopy will be performed at 6 weeks.

After 6 weeks, patients will once again undergo bronchoscopy with BAL/biopsies. Cytokine protein arrays will be repeated. Comparisons will then be made intra-group before and after therapy. Additional comparisons of inflammation and bronchial hyper-responsiveness will be made between groups. Randomization will allow the investigators to control for any changes in cytokine patterns due to seasonal affect (if both groups reduce the concentration of Interleukin-5 in a similar pattern, this is more likely seasonal than due to acid suppression).

Primary outcome will include change in cellular infiltration in the bronch specimens of lymphocytes. Secondary outcome will include RNA expression changes of tumor necrosis factor (TNF) alpha from BAL samples.

ELIGIBILITY:
Inclusion Criteria:

1. chronic cough consistent with bronchoreactivity
2. Gastroesophageal reflux

Exclusion Criteria:

1. Severe asthmatics who have been hospitalized within the last 6 months or who have required oral steroid use within the last 4 weeks
2. Severe coronary artery disease
3. Cigarette/cigar smoking within the last 6 months
4. Documented allergies affecting the respiratory system
5. Subjects with contraindications to pH/impedance probe

   1. Hemophilia
   2. Septal deviation
6. Subjects with contraindications to bronchoscopy as outlined by the American Thoracic Society Guidelines
7. Anticoagulation
8. Pregnancy
9. Incarcerated patients
10. Current oral steroid use (may suppress levels of inflammation)
11. Upper respiratory infection within the last 2 weeks
12. Ongoing acid suppression with a proton pump inhibitor, however, patients may be included if they have discontinued their proton pump inhibitor within the last 1 month with stable asthma symptoms as defined by stable utilization of inhaled steroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Peterson, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: in clinics over 18 month period
Pre-assignment Details: washout after lansoprazole or placebo given
Groups:
- Lansoprazole: lansoprazole : 30 mg of lansoprazole twice daily for 6 weeks
- Placebo: placebo comparator to lansoprazole, 30 mg, twice a day for 6 weeks
Period: Overall Study
Arm/Group | Lansoprazole | Placebo
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: placebo comparator to lansoprazole 30 mg twice daily for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Lansoprazole | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Full Range); unit: years] | 40 [20 to 57] | 43 [26 to 62] | 41 [20 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Lymphocyte Count
Description: Change in mean lymphocyte count in bronchus intermedius biopsies between lansoprazole and placebo groups, measured in lymphocytes per square millimeter. Overall mean differences were compared (post-intervention mean lymphocyte count minus pre-intervention mean lymphocyte count) between the two intervention groups.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: Lymphocytes per square millimeter
Groups:
- Lansoprazole: lansoprazole: 30 mg lansoprazole twice daily for 6 weeks
Arm/Group | Lansoprazole | Placebo
Number analyzed (Participants) | 8 | 9
Lymphocytes per square millimeter | -57 (10) | -3 (2)
Statistical Analysis 1: Comparison: Lansoprazole vs Placebo; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Log Change in Tumor Necrosis Factor (TNF) Alpha Measurement
Description: Change in TNF alpha cytokine expression from bronchoalveolar lavage aspirate samples between lansoprazole and placebo groups, measured in log picograms per milliliter (log (pg/mL)) units, pre- and post-intervention.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: log (pg/mL)
Arm/Group | Lansoprazole | Placebo
Number analyzed (Participants) | 8 | 9
log (pg/mL) | 0.4 [-1.4 to 1.5] | 2.0 [-1.6 to 5.6]
Statistical Analysis 1: Comparison: Lansoprazole vs Placebo; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Lansoprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

LIMITATIONS AND CAVEATS:
Questionnaires were not assessed as many of them were incomplete. Drop out occurred due to incomplete tissues Early termination: the total number of participants could not be enrolled in a timely manner..

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No